CLINICAL TRIAL: NCT06014697
Title: The Value of Optical Coherence Tomography in Discrimination Between the Presence and Absence of Invasion in Clinical Actinic Keratosis
Brief Title: OCT and Invasion in Cutaneous Skin Lesions
Status: Completed | Type: Observational
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2023-3735
Record Dates: First submitted 2023-08-15; First posted 2023-08-28 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-03

CONDITIONS: Cutaneous Squamous Cell Carcinoma; Bowen's Disease; Actinic Keratoses; Keratosis, Actinic; Diagnosis
Keywords: Optical coherence tomography; Invasion; Diagnostic device; Non-invasive
MeSH Terms: conditions — Bowen's Disease; Keratosis, Actinic; Disease | interventions — Tomography, Optical Coherence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Non-invasive lesion: Lesion with histological confirmation of a actinic keratosis or Bowens disease (non-invasive lesions).
  Interventions: Diagnostic Test: Optical Coherence Tomography; Other: Clinical assessment
- Invasive lesion: Lesion with histological confirmation of a squamous cell carcinoma (invasive lesions).
  Interventions: Diagnostic Test: Optical Coherence Tomography; Other: Clinical assessment

INTERVENTIONS:
Diagnostic Test: Optical Coherence Tomography — Assessment of the lesion with a non-invasive OCT scan according to a confidence scale (5-point Likert scale: 1 Definitely not invasive, 2 Probably not invasive, 3 Unknown invasive or non-invasive, 4 Probably invasive, 5 Definitely invasive)
  Other Names: OCT
Other: Clinical assessment — Clinical assessment of the lesion by a dermatologist according to a confidence scale (5-point Likert scale: 1 Definitely not invasive, 2 Probably not invasive, 3 Unknown invasive or non-invasive, 4 Probably invasive, 5 Definitely invasive)

SUMMARY:
The increasing incidence of actinic keratosis (AK), morbus Bowen (MB) and cutaneous squamous cell carcinoma (cSCC), the patients with often multiple lesions and the disadvantages of invasive diagnostics show the need for an accurate non-invasive diagnostic tool for the determination of invasive growth in AK and MB.

Optical coherence tomography (OCT) is a non-invasive scanner creating cross-sectional images of the skin, to a depth of 1-1,5 mm based on light waves. Until now, OCT has been proposed as non-invasive diagnostic tool for basal cell carcinomas. Although the diagnostic value of OCT for detection and sub-typing of basal cell carcinomas has already been demonstrated, it is unclear whether OCT can discriminate between invasive and non-invasive lesions (AK, MB and cSCCs). There are some studies that describe OCT characteristics of AK, MB and cSCCs, however, these characteristics have a lot of overlap (8-13). To date there are no clearly distinctive OCT features to distinguish between AK, MB and cSCCs. This study aims to investigate the value of OCT in discriminating between the presence and absence of invasion in lesions with clinical suspicion for invasion.

Two experienced OCT-assessors will evaluate the OCT scans independently. The OCT assessors are blinded to the histological diagnosis of the lesions (invasive or non-invasive), which is used as golden standard.

A 5-point Likert scale is used for OCT assessment.

1. Definitely not invasive
2. Probably not invasive
3. Unknown, probably invasive/probably not invasive
4. Probably invasive
5. Definitely invasive

In addition to completing the Likert-scale, assessors are asked to describe the presence/absence of predefined OCT characteristics (a.o. hyperkeratosis and the presence of the dermo-epidermal junction)

In case of disagreement between the independent assessors, the OCT scan will be re-assessed in a consensus meeting.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are included in a previous study on OCT, with written informed consent to use their data regarding OCT.
* Patients who retrospectively had an OCT scan for their skin lesion
* With a histological confirmed actinic keratosis, bowens disease or cutaneous squamous cell carcinoma of the skin
* with a differential diagnosis of a invasive lesion (cutaneous squamous cell carcinoma) and a non-invasive lesion (bowens disease or actinic keratosis).

Exclusion Criteria:

* patients who waived informed consent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patient with a histologically confirmed actinic keratosis, bowens disease or cutaneous squamous cell carcinoma, with a clinical differential diagnosis of actinic keratosis and/or bowens disease and cutaneous squamous cell carcinoma, included in a previous study. All patients retrospectively had a OCT scan.
Sampling Method: Non-Probability Sample
Enrollment: 71 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2024-08-01 (Actual)

PRIMARY OUTCOMES:
Sensitivity | Through study completion, an average of 6 months
  Sensitivity of OCT to detect invasion
Specificity | Through study completion, an average of 6 months
  Specificity of OCT in determining the presence/absence of invasion

SECONDARY OUTCOMES:
Negative predictive value | Through study completion, an average of 6 months
  Negative predictive value of OCT in determining the presence/absence of invasion
Positive predictive value | Through study completion, an average of 6 months
  Positive predictive value of OCT in determining the presence/absence of invasion
Area under the curve | Through study completion, an average of 6 months
  Area under the curve for OCT in determining the presence/absence of invasion
Sensitivity of OCT features | Through study completion, an average of 6 months
  Sensitivity for specific OCT-features characteristic for the presence/absence of invasion, such as presence/absence of the dermo-epidermal junction or presence/absence of hyperkeratosis.
Difference OCT and clinical practice | Through study completion, an average of 6 months
  Difference in diagnostic parameters (sensitivity, specificity and area under the curve) between OCT and clinical practice (clinical assessment).
Specificity of OCT features | Through study completion, an average of 6 months
  Specificity for specific OCT-features characteristic for the presence/absence of invasion, such as presence/absence of the dermo-epidermal junction or presence/absence of hyperkeratosis.
Positive predictive value of OCT features | Through study completion, an average of 6 months
  Positive predictive value for specific OCT-features characteristic for the presence/absence of invasion, such as presence/absence of the dermo-epidermal junction or presence/absence of hyperkeratosis.
Negative predictive value of OCT features | Through study completion, an average of 6 months
  Negative predictive value for specific OCT-features characteristic for the presence/absence of invasion, such as presence/absence of the dermo-epidermal junction or presence/absence of hyperkeratosis.
Area under the curve for OCT features | Through study completion, an average of 6 months
  Area under the curve for specific OCT-features characteristic for the presence/absence of invasion, such as presence/absence of the dermo-epidermal junction or presence/absence of hyperkeratosis.

CONTACTS AND LOCATIONS:
Overall Officials: K Mosterd, MD, PhD, Principal Investigator — Maastricht University Medical Center
Locations (1):
- Maastricht University Medical Center+, Maastricht, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Stratigos AJ, Garbe C, Dessinioti C, Lebbe C, Bataille V, Bastholt L, Dreno B, Fargnoli MC, Forsea AM, Frenard C, Harwood CAlpha, Hauschild A, Hoeller C, Kandolf-Sekulovic L, Kaufmann R, Kelleners-Smeets NW, Malvehy J, Del Marmol V, Middleton MR, Moreno-Ramirez D, Pellecani G, Peris K, Saiag P, van den Beuken-van Everdingen MHJ, Vieira R, Zalaudek I, Eggermont AMM, Grob JJ; European Dermatology Forum (EDF), the European Association of Dermato-Oncology (EADO) and the European Organization for Research and Treatment of Cancer (EORTC). European interdisciplinary guideline on invasive squamous cell carcinoma of the skin: Part 1. epidemiology, diagnostics and prevention. Eur J Cancer. 2020 Mar;128:60-82. doi: 10.1016/j.ejca.2020.01.007. Epub 2020 Feb 26. PMID 32113941
- [Background] Hollestein LM, de Vries E, Nijsten T. Trends of cutaneous squamous cell carcinoma in the Netherlands: increased incidence rates, but stable relative survival and mortality 1989-2008. Eur J Cancer. 2012 Sep;48(13):2046-53. doi: 10.1016/j.ejca.2012.01.003. Epub 2012 Feb 16. PMID 22342554
- [Background] Lomas A, Leonardi-Bee J, Bath-Hextall F. A systematic review of worldwide incidence of nonmelanoma skin cancer. Br J Dermatol. 2012 May;166(5):1069-80. doi: 10.1111/j.1365-2133.2012.10830.x. PMID 22251204
- [Background] Sinx KAE, van Loo E, Tonk EHJ, Kelleners-Smeets NWJ, Winnepenninckx VJL, Nelemans PJ, Mosterd K. Optical Coherence Tomography for Noninvasive Diagnosis and Subtyping of Basal Cell Carcinoma: A Prospective Cohort Study. J Invest Dermatol. 2020 Oct;140(10):1962-1967. doi: 10.1016/j.jid.2020.01.034. Epub 2020 Mar 6. PMID 32147505
- [Background] Moy RL. Clinical presentation of actinic keratoses and squamous cell carcinoma. J Am Acad Dermatol. 2000 Jan;42(1 Pt 2):8-10. doi: 10.1067/mjd.2000.103343. PMID 10607350
- [Background] Ahmady S, Jansen MHE, Nelemans PJ, Kessels JPHM, Arits AHMM, de Rooij MJM, Essers BAB, Quaedvlieg PJF, Kelleners-Smeets NWJ, Mosterd K. Risk of Invasive Cutaneous Squamous Cell Carcinoma After Different Treatments for Actinic Keratosis: A Secondary Analysis of a Randomized Clinical Trial. JAMA Dermatol. 2022 Jun 1;158(6):634-640. doi: 10.1001/jamadermatol.2022.1034. PMID 35475852
- [Background] Levine A, Wang K, Markowitz O. Optical Coherence Tomography in the Diagnosis of Skin Cancer. Dermatol Clin. 2017 Oct;35(4):465-488. doi: 10.1016/j.det.2017.06.008. Epub 2017 Aug 9. PMID 28886803
- [Background] Sattler E, Kastle R, Welzel J. Optical coherence tomography in dermatology. J Biomed Opt. 2013 Jun;18(6):061224. doi: 10.1117/1.JBO.18.6.061224. PMID 23314617
- [Background] Boone MA, Marneffe A, Suppa M, Miyamoto M, Alarcon I, Hofmann-Wellenhof R, Malvehy J, Pellacani G, Del Marmol V. High-definition optical coherence tomography algorithm for the discrimination of actinic keratosis from normal skin and from squamous cell carcinoma. J Eur Acad Dermatol Venereol. 2015 Aug;29(8):1606-15. doi: 10.1111/jdv.12954. Epub 2015 Feb 5. PMID 25656269
- [Background] Marneffe A, Suppa M, Miyamoto M, Del Marmol V, Boone M. Validation of a diagnostic algorithm for the discrimination of actinic keratosis from normal skin and squamous cell carcinoma by means of high-definition optical coherence tomography. Exp Dermatol. 2016 Sep;25(9):684-7. doi: 10.1111/exd.13036. PMID 27095632
- [Background] Friis KBE, Themstrup L, Jemec GBE. Optical coherence tomography in the diagnosis of actinic keratosis-A systematic review. Photodiagnosis Photodyn Ther. 2017 Jun;18:98-104. doi: 10.1016/j.pdpdt.2017.02.003. Epub 2017 Feb 7. PMID 28188920
- See also: VivoSight OCT Education Centre. VivoSight. 2022. — https://www.vivosightatlas.com/